CLINICAL TRIAL: NCT03006029
Title: A Phase 1b Multiple Dose Escalation Study of TAB08 in Patients With Advanced Solid Neoplasms
Brief Title: Dose Escalation Study of TAB08 in Patients With Advanced Solid Neoplasms
Acronym: TAB08
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theramab LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAB08-ONC-01
Record Dates: First submitted 2016-11-29; First posted 2016-12-30 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Solid Tumors
MeSH Terms: interventions — TGN-1412

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAB08( Theralizumab) (Experimental): TAB08 will be administered i.v. over 1 hour weekly for 3 weeks followed by 3 weeks of no treatment; with 6 weeks interval between start of each treatment cycle.
  Interventions: Drug: TAB08

INTERVENTIONS:
Drug: TAB08 — The initial dose of TAB08 will be 1 µg/kg TAB08 will be administered i.v. over 1 hour weekly for 3 weeks followed by 3 weeks of no treatment; with 6 weeks interval between start of each treatment cycle.
  Other Names: Theralizumab

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose of TAB08 when administered intravenously (i.v.) to patients with advanced solid malignancies.

DETAILED DESCRIPTION:
This is an open-label, multi-center, sequential groups, dose escalation study of TAB08 in patients with metastatic or unresectable advanced solid malignancies. The study will consist of 2 parts: a dose-escalation part with a standard "3+3" design, followed by a dose-expansion part once the maximum tolerated dose (MTD) has been determined.

Patients must have documented recurrent or refractory solid tumors; patients enrolled in the dose-expansion part of the trial must have least one lesion that may qualify as a target lesion based on the RECIST 1.1 criteria. Following the provision of signed informed consent, patients will be screened for entry into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects or their authorized representatives must be able to provide written informed consent.
2. Subjects must have histological or cytological evidence of a solid neoplasm for which standard therapy has failed or does not exist or is not available for patient due to any reason.
3. Subjects enrolled in the expansion cohort must have at least one measurable evaluable lesion.
4. Subjects must have ECOG (Eastern Cooperation Oncology Group) performance status of 0 or 1.
5. Subjects must be ≥ 18 years of age.
6. Subjects must have adequate organ function, as defined by the following criteria:

   * Absolute neutrophil count (ANC) > 1,500/µL.
   * Platelet count > 75,000/µL.
   * Hemoglobin (Hb) > 8.0 g/dL.
   * Serum creatinine of < 1.5 x upper limit of normal (ULN) or a calculated Glomerular Filtration Rate of >40 mL/min/1.73m2.
   * Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN (< 5 x ULN for subjects with known liver metastases).
7. At least 2 weeks or at least 5 half-lives must have elapsed since prior treatment with chemotherapy, targeted therapy, radiotherapy, immunotherapy, or investigational anti-cancer therapy prior to study drug administration. The maximum washout period will not exceed 4 weeks. .
8. Subjects must have recovered from the effects of any prior surgery, radiotherapy, localized therapy, or systemic therapy to Grade 1 or lower (except alopecia or anemia - Grade 2 permitted).
9. Subjects have a life expectancy ≥ 3 months at study entry.
10. Women of childbearing potential and men with partners of childbearing potential must agree to abstain from sexual intercourse or use an effective form of contraception.

Exclusion Criteria:

1. Subjects with an uncontrolled concurrent illness, including, but not limited to the following: ongoing active infection requiring systemic treatment; uncontrolled endocrine disease; diabetes mellitus or chronic obstructive pulmonary disease (COPD) requiring hospitalization within the preceding 6 months.
2. Subjects with uncontrolled arterial hypertension, heart failure by New York Heart Association (NYHA) Class 3 or 4, left ventricular ejection fraction (LVEF) < 50% by echocardiography, myocardial infarction, acute coronary syndrome and/or QT prolongations within the preceding 6 months or history of cerebrovascular accidents including episodes of transient ischemic attacks.
3. Subjects with altered mental status or psychiatric illness or social circumstances that would limit compliance with the study requirements and/or obscure the results.
4. Immunocompromised subjects, e.g., subjects known to be infected with human immunodeficiency virus (HIV) by medical history, and subjects with active hepatitis A, B, or C by medical history.
5. Subjects having untreated or symptomatic brain metastasis, or subjects with leptomeningeal disease. (Subjects with treated metastases, who are off corticosteroids and who are neurologically stable for at least 2 months may participate in the trial.)
6. A history of major surgery within 28 days prior to the first dose of study drug.
7. Subjects with history of other malignancies within the preceding 5 years (except for subjects with non-melanoma skin cancers, cervical intra-epithelial neoplasia, prostate cancer Gleason ≤ 6 and Prostate Specific Antigen (PSA) < 10 ng/mL, radically excised lobular breast carcinoma in situ or ductal breast carcinoma in situ ≤ 15 mm) unless they have undergone potentially curative therapy and have had no evidence of disease for 3 years (ie, 5 years since diagnosis, no treatment or symptoms of disease for the last 3 years).
8. Women who are pregnant or nursing.
9. Subjects with any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the opinion of the investigator, contraindicates use of the investigational drug, or may render the subject as excessively high risk for treatment complications.
10. Subjects with any other condition as determined by medical history, including substance abuse that, in the opinion of the investigator, would render the subject unable to cooperate in the trial or place the subject at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Number of cases of the Dose-limiting toxicity (DLT) | DLT assessment will be performed within first 2 weeks of treatment

SECONDARY OUTCOMES:
Adverse events (including local reactions) frequency, seriousness and severity | Through study completion, not less than 8 weeks
TAB08 concentrations in peripheral blood | First 4 weeks of TAB08 administration
Tumor response to TAB08 according to immune-related Response Criteria in Solid Tumors (irRECIST) | Through study completion, not less than 12 weeks
Change of T-lymphocytes subsets in absolute count (number of cells per mL) in peripheral blood at designated timepoints comparing to Baseline. | Through study completion, not less than 8 weeks
Change of T-lymphocytes subsets in percent in peripheral blood at designated timepoints comparing to Baseline. | Through study completion, not less than 8 weeks
Change of cytokines concentrations (in micrograms/mL) in peripheral blood at designated timepoints comparing to Baseline. | Through study completion, not less than 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniil G Nemenov, MD, Study Director — Theramab LLC
Locations (1):
- GBU Ryazanskoy Oblasti "Oblastnoy klinicheckiy oncologicheskiy dispanser", Ryazan, Russia

IPD SHARING:
Plan to Share IPD: No